CLINICAL TRIAL: NCT07180888
Title: Study of Diastolic Dysfunction in ESKD in Hemodialysis Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaaeldien Hamed Hamada, egypt sohag, Sohag University
Other Study IDs: soh-med-25-7-21MS
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; ESKD; Hemodialysis Patients
Keywords: echocardiography; dialysis patients
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — diastolic dysfunction in ESKD in hemodialysis by echocardiography
Diagnostic Test: Echocardiographic assessment of diastolic dysfunction — non invasive transthoracic echocardiography including doppler and tissue doppler imaging will be used to assess left ventricular diastolic dysfunction parameters in hemodialysis patient

SUMMARY:
To Asses the prevalence , pattern , and severity of diastolic dysfunction in patients ESKD undergoing regular dialysis and to investigate its correlation with clinical parameters dialysis-related factors and echocardiographic findings

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years not diagnosed by MI able and willing to provide informed consent

Exclusion Criteria:

previous MI arrythmia CHF

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patient with on hemodialysis with diastolic heart failure in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
diastolic dysfunction in ESKD in hemodialysis patient | 4 months
  diastolic dysfunction by transthoracic Echocardiography in hemodialysis patients

IPD SHARING:
Plan to Share IPD: No
fot save patients privacy